CLINICAL TRIAL: NCT03332680
Title: A Randomised Controlled Trial Assessing the Effectiveness of EmbryoGlue® as an Embryo Transfer Medium in IVF Treatment Cycles
Brief Title: EmbryoGlue as an Embryo Transfer Medium
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Oxford (Other)
Collaborators: Oxford Fertility Limited, United Kingdom (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NDOG-17/NW/0272
Record Dates: First submitted 2017-05-17; First posted 2017-11-06 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: This study is a positive control study with a single site two arm parallel design
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: In terms of blinding, the physician and/or nurses as well as the patients will be blinded and will not know what arm of the study the participant has been allocated too. The embryologists however will be unblinded (as they provide intervention and will have to be aware).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EmbryoGlue® (laboratory culture medium) (Experimental): laboratory culture medium
  laboratory embryo culture medium, embryos are placed in this media prior to transfer into uterus via embryo transfer procedure to facilitate IVF. EmbryoGlue contains Hyaluronic acid.
  Interventions: Biological: EmbryoGlue® (laboratory culture medium)
- Standard control medium (Active Comparator): laboratory culture medium
  In standard procedure embryos are placed in a media prior to transfer into uterus via embryo transfer procedure to facilitate IVF.
  Interventions: Biological: Standard control medium

INTERVENTIONS:
Biological: EmbryoGlue® (laboratory culture medium) — Embryos placed in this medium prior to transfer
  Other Names: EmbryoGlue
  Arms: EmbryoGlue® (laboratory culture medium)
Biological: Standard control medium — Embryos placed in this medium prior to transfer
  Arms: Standard control medium

SUMMARY:
In Vitro Fertilisation (IVF) is an increasingly common treatment for infertility. Clinics which offer IVF are continuously trying to improve their success rates, measured by the numbers of IVF cycles which result in the birth of a live baby.

One factor which is thought to have contributed to the success of IVF is the improvements in the embryo culture media, that is, the fluid in which the embryo resides in the laboratory before being replaced into a woman's womb. This trial seeks to identify if IVF cycles in which a particular culture media called EmbryoGlue is used have better results when compared to IVF cycles in which a conventional embryo transfer media is used.

ELIGIBILITY:
Inclusion Criteria:

• Couples having embryo transfer for fertility treatment

Exclusion Criteria:

* Cycles in which elective freezing of all embryos is clinically indicated (e.g. severe risk of OHSS, biopsy patients)
* Use of donor gametes
* Having endometrial scratch technique this cycle
* Concurrent participation in clinical trial(s)
* Previously randomised to this study
* Planned self-fund of EmbryoGlue as transfer media

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 730 (Estimated)
Dates: Start 2017-06-16 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
Live Birth Rate | outcome data up to 9 months after intervention

SECONDARY OUTCOMES:
Implantation rate | outcome data up to 9 months after intervention
Clinical pregnancy rates, | outcome data up to 9 months after intervention
Adverse IVF events. | outcome data up to 9 months after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford Fertility, Oxford, United Kingdom